CLINICAL TRIAL: NCT05636592
Title: Statin Combined With PD-1/PD-L1 Inhibitors in Treating NSCLC
Brief Title: Combined Statin and PD-1/PD-L1 Inhibitors in Treating Non-small Cell Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: K2022145
Record Dates: First submitted 2022-11-18; First posted 2022-12-05 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard programme group: Standard programme group, immunotherapy alone
- controlled programme group: controlled programme group, statin combined with immunotherapy
  Interventions: Drug: immunotherapy

INTERVENTIONS:
Drug: immunotherapy — statin combined with immunotherapy
  Groups: controlled programme group

SUMMARY:
This prospective observational study was designed to evaluate the safety and efficacy of PD-1/PD-L1 inhibitors in combination with statins compared with treatment with PD-1/PD-L1 inhibitors alone in advanced NSCLC patients. Participants will receive either immunotherapy + statin or immunotherapy until progressive disease (PD) as assessed by the investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). Treatment can be continued until persistent radiographic PD or symptomatic deterioration.

DETAILED DESCRIPTION:
Statin is an inhibitor of 3-hydroxy-3-methylglutaryl-coenzyme A (CoA) reductase (HMGCR), the rate-limiting enzyme of the mevalonate (MVA) pathway for the cholesterol biosynthesis. Statins reportedly target the immune microenvironment through cytokines or chemokines and immune checkpoints. In a B16 melanoma lung metastatic model, statin lowers PD-1 expression in CD8+ T cells and effectively restores antitumor activity. In colorectal cancers model, simvastatin acts as a potential therapeutic drug for immunotherapy, which suppresses lncRNA SNHG29-mediated YAP activation and promotes anti-tumor immunity by inhibiting PD-L1 expression. Some retrospective observational studies have reported that baseline statin use was associated with improved clinical activity of PD-1/PD-L1 inhibitors in non-small cell lung cancer (NSCLC) patients. These findings support the adjuvant role of statins combined with immunotherapy. Statin therapy may be a combination tool for cancer immunotherapy in patients with NSCLC. Data from already completed clinical trials are not always supportive. These findings should be validated in further prospective studies with larger sample sizes. More clinical trials are needed to explore the right drug type, dose, frequency, duration, and suitable participator. Thus, this prospective observational study was designed to evaluate the safety and efficacy of PD-1/PD-L1 inhibitors in combination with statins compared with treatment with PD-1/PD-L1 inhibitors alone in advanced NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology or hemology diagnostics of phase IIIB or IV (AJCC Version 8) NSCLC that cannot be surgicalor-able or radiotherapy
* Not applicable to EGFR/ALK/ROS1 targeted therapy
* Within 4 weeks prior to randomization, at least one measurable target lesions assessed by irRC in accordance with RECIST 1.1 requirements
* Patients have never received PD-1/PD-L1/CTLA-4 inhibitors treatment throughout the body for phase IIIB or IV NSCLC
* Patient have indications for statins
* The ECOG PS score for 7 days prior to the first drug use of the study drug was 0 or 1
* The expected lifetime is more than 12 weeks
* The main organ function sits well, i.e. meets the following criteria (no blood transfusion, albumin, recombinant human platelet production or Colony-stimulating factor (CSF) treatment within 14 days prior to the first drug use in this study)

Exclusion Criteria:

* Within 5 years or at the same time, there are other active malignancies. Cured limited tumors, such as skin base cell carcinoma, skin squamous carcinoma, superficial bladder cancer, prostate in situ cancer, cervical in situ cancer, etc. can be included in the group
* Currently participating in interventional clinical research treatment, or received other research drugs or used research devices within 4 weeks before the first administration
* Active autoimmune diseases requiring systemic treatment (such as the use of disease relieving drugs, glucocorticoids or immunosuppressants) occurred within 2 years before the first administration
* The study was receiving systemic glucocorticoid treatment (excluding local glucocorticoids by nasal spray, inhalation or other means) or any other form of immunosuppressive therapy within 7 days before the first administration; Note: It is allowed to use glucocorticoid with physiological dose (prednisone ≤ 10mg/day or equivalent)
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
* According to the instructions of statins, there are contraindications to the use of statins
* People who are allergic to any component of the drug
* People with multiple factors affecting oral medicine (such as inability to swallow, gastrointestinal resection, significant digestive system diseases that may interfere with absorption, metabolism or excretion, such as chronic diarrhea or intestinal obstruction)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to indications of statins, the enrolled people are divided into statin group and non-statin group.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate | three years
  Refers to the proportion of patients whose tumor shrinkage reaches a certain amount and remains for a certain period of time, including CR + PR cases
progression-free survival | three years
  Patients with oncological diseases have a period of time from the start of treatment to the observation of disease progression or death due to any cause

SECONDARY OUTCOMES:
overall survival | five years
  The time from randomization to death due to any cause. For subjects who have been lost to follow-up before death, the time of the last follow-up is usually calculated as the time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, PhD, Study Chair — The Fourth Affiliated Hospital of Zhejiang University
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided